CLINICAL TRIAL: NCT03382366
Title: Sarcopenia and Risk of Fall in Elder Post-menopausal Osteoporotic Women: a Pilot Study
Brief Title: Sarcopenia and Risk of Fall in Osteoporotic Postmenopausal Women
Acronym: Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Sarcopenia
Record Dates: First submitted 2017-12-04; First posted 2017-12-22 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Sarcopenia; Falls Patient; Osteoporosis, Postmenopausal
Keywords: Sarcopenia; Risk of fall; Osteoporosis; Muscle; DXA; MR; Muscle metabolism
MeSH Terms: conditions — Sarcopenia; Osteoporosis, Postmenopausal; Osteoporosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sarcopenic Group (Other): This group is composed by 20 osteoporotic postmenopausal women, previously (pre-recruitment) classified as "sarcopenic" by the DXA.
  This group will undergo the same evaluations/intervention of the second group.
  Interventions: Diagnostic Test: Blood sampling, risk of fall evaluation, and MR acquisition.
- Non-sarcopenic Group (Other): This group is composed by 20 osteoporotic postmenopausal women, previously (pre-recruitment) classified as "non-sarcopenic" by the DXA.
  This group will undergo the same evaluations/intervention of the first group.
  Interventions: Diagnostic Test: Blood sampling, risk of fall evaluation, and MR acquisition.

INTERVENTIONS:
Diagnostic Test: Blood sampling, risk of fall evaluation, and MR acquisition. — Data will be collected on 1) bone/muscle metabolism through blood sampling, 2) risk of fall through OAK device; 3) muscle quality through MR acquisition.

SUMMARY:
The main scope of the present pilot study is to evaluate the possible association between the status of sarcopenia and the risk of fall in osteoporotic postmenopausal women. Forty osteoporotic postmenopausal women, previously (pre-recruitment) classified by DXA in 20 sarcopenic and 20 non-sarcopenic subjects, will be recruited. The investigators will collect data on: 1) bone (vitamin D) and muscle (myokines) metabolisms through blood sampling; 2) Risk of fall by the OAK device produced by Khymeia; 3) thigh muscle quality through MR.

DETAILED DESCRIPTION:
A grave change associated with human ageing is progressive decline in skeletal muscle mass, a downward spiral that may lead to decreased strength and functionality. The term 'sarcopenia' (Greek 'sarx' or flesh + 'penia' or loss) has been proposed to describe this age-related decrease of muscle mass. Sarcopenia represents an impaired state of health with increased risk of falls and fractures, impaired ability to perform activities of daily living, and loss of independence. The imaging technologies used to detect loss of skeletal muscle mass in sarcopenia include: dual X-ray absorptiometry (DXA), magnetic resonance imaging (MR), computed tomography, peripheral quantitative computed tomography, and ultrasound.

The main scope of the present pilot study is to evaluate the possible association between the status of sarcopenia and the risk of fall in osteoporotic postmenopausal women. Forty osteoporotic postmenopausal women, previously (pre-recruitment) classified by DXA in 20 sarcopenic and 20 non-sarcopenic subjects, will be recruited. Data will be collected on: 1) bone (vitamin D) and muscle (myokines) metabolisms through blood sampling; 2) Risk of fall by the OAK device produced by Khymeia; 3) thigh muscle quality through MR.

A secondary outcome is to evaluate the differences in bone and muscle metabolism, risk of fall, and muscle quality between sarcopenic and non-sarcopenic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Female.
* Aged over 60 yo.
* Classified as osteoporotic with t-score = or < -2,5 evaluated by DXA.
* Autonomous walking.
* Signed informed consent.

Exclusion Criteria:

* Male.
* Aged under 60 yo.
* Psychiatric disorders.
* Neurological pathologies.
* Endocrine disorders.
* Active cigarettes smoke.
* Recent bone fractures (6 months)
* Surgical treatments for orthopedic pathologies (6 months).
* Pacemaker carrier.
* Use of drugs influencing bone metabolism or limiting physical function.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-29 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Association between sarcopenia, meant as the percentage of fat fraction of the thigh muscle evaluated by RM, and risk of fall evaluated through the OAK device. | 2 days.
  The fat fraction of the thigh muscle is obtained by RM and expressed in percentage (%) of fat on muscle.
  The risk of fall will be derived by the final score of the OAK device system. The score range is 0-24. Higher scores represent lower risk of falls.
Association between sarcopenia, meant as the Appensicular Skeletal Muscle Mass Index (ASMMI) obtained by DXA, and risk of fall evaluated through the OAK device. | 2 days.
  ASMMI is obtained by DXA and calculated with the following formula: (total grams of lean muscle mass of left and right lower and upper limbs)/height*height, expressed in meters.
  The risk of fall will be derived by the final score of the OAK device system. The score range is 0-24. Higher scores represent lower risk of falls.

SECONDARY OUTCOMES:
Comparison of the fat fraction of the thigh muscle, obtained by RM, between sarcopenic and non-sarcopenic subjects. | 2 days.
  Compare the data collected on the fat fraction of the thigh muscle, obtained by RM and expressed in percentage of fat on muscle, between sarcopenic and non-sarcopenic osteoporotic women.
Comparison of risk of fall, evaluated with the use of the OAK device, between sarcopenic and non-sarcopenic subjects. | 2 days.
  The OAK device is an innovative technologic system, based on virtual reality, for the assessment and prevention of risk of fall in the elderly. The OAK device comprises (i) two stabilometric platforms that register the Center of Pressure (CoP) of each limb, (ii) four antennas, responsible for the low intensity magnetic field generation into which the patient will move, (iii) three bars able to detect the body weight loaded by the patient during the exercise accomplishment and (iv) a monitor, through which the patient is able to hear and see the exercises proposed. The subject will be set up with a belt, two gloves and two wrappers, containing passive magnetic sensors which can register subject's motions in real time thanks to the magnetic field generated by the antennas.
  The fall risk assessment will last about 10 minutes and it will be performed before and after the exercise training. A score regarding the fall risk (low, medium or high risk) of the subject will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Lourenco RA, Perez-Zepeda M, Gutierrez-Robledo L, Garcia-Garcia FJ, Rodriguez Manas L. Performance of the European Working Group on Sarcopenia in Older People algorithm in screening older adults for muscle mass assessment. Age Ageing. 2015 Mar;44(2):334-8. doi: 10.1093/ageing/afu192. Epub 2014 Dec 23. PMID 25539836
- [Background] Sergi G, Trevisan C, Veronese N, Lucato P, Manzato E. Imaging of sarcopenia. Eur J Radiol. 2016 Aug;85(8):1519-24. doi: 10.1016/j.ejrad.2016.04.009. Epub 2016 Apr 14. PMID 27117135
- [Background] Tosato M, Marzetti E, Cesari M, Savera G, Miller RR, Bernabei R, Landi F, Calvani R. Measurement of muscle mass in sarcopenia: from imaging to biochemical markers. Aging Clin Exp Res. 2017 Feb;29(1):19-27. doi: 10.1007/s40520-016-0717-0. Epub 2017 Feb 7. PMID 28176249
- [Background] Rubbieri G, Mossello E, Di Bari M. Techniques for the diagnosis of sarcopenia. Clin Cases Miner Bone Metab. 2014 Sep;11(3):181-4. PMID 25568650
- [Background] Baumgartner RN, Koehler KM, Gallagher D, Romero L, Heymsfield SB, Ross RR, Garry PJ, Lindeman RD. Epidemiology of sarcopenia among the elderly in New Mexico. Am J Epidemiol. 1998 Apr 15;147(8):755-63. doi: 10.1093/oxfordjournals.aje.a009520. PMID 9554417
- [Background] Roubenoff R, Hughes VA. Sarcopenia: current concepts. J Gerontol A Biol Sci Med Sci. 2000 Dec;55(12):M716-24. doi: 10.1093/gerona/55.12.m716. PMID 11129393
- [Background] Cummings-Vaughn LA, Gammack JK. Falls, osteoporosis, and hip fractures. Med Clin North Am. 2011 May;95(3):495-506, x. doi: 10.1016/j.mcna.2011.03.003. PMID 21549874
- [Background] Tyson SF, Connell LA. How to measure balance in clinical practice. A systematic review of the psychometrics and clinical utility of measures of balance activity for neurological conditions. Clin Rehabil. 2009 Sep;23(9):824-40. doi: 10.1177/0269215509335018. Epub 2009 Aug 5. PMID 19656816
- [Background] Dixon WT. Simple proton spectroscopic imaging. Radiology. 1984 Oct;153(1):189-94. doi: 10.1148/radiology.153.1.6089263.